CLINICAL TRIAL: NCT04494334
Title: Development of Airway Absorption Sampling Methods for Biomarker Assessment in Probable Idiopathic Pulmonary Fibrosis (IPF) Patients
Brief Title: Development of Airway Absorption Sampling Methods
Acronym: FIBRO-SAM
Status: Withdrawn | Type: Observational
Why Stopped: Study terminated by funder- terminated before CCC and recruitment- no recruitment and no data collection
Sponsor: Imperial College London (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19SM5398; 239911 (Other: IRAS)
Record Dates: First submitted 2020-06-09; First posted 2020-07-31 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Idiopathic Pulmonary Fibrosis; Sarcoidosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Sarcoidosis | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: These will be age matched healthy volunteers (n=15) who will not undergo bronchoscopy
- Probable Idiopathic Pulmonary Fibrosis: Patients with probable IPF, who will be having bronchoscopy as part of their clinical diagnostic work up
  Interventions: Procedure: Bronchoscopy for Probable Idiopathic Pulmonary Fibrosis and Sarcoidosis
- Sarcoidosis,: Patients with sarcoidosis who will be having bronchoscopy as part of their clinical diagnostic work up
  Interventions: Procedure: Bronchoscopy for Probable Idiopathic Pulmonary Fibrosis and Sarcoidosis

INTERVENTIONS:
Procedure: Bronchoscopy for Probable Idiopathic Pulmonary Fibrosis and Sarcoidosis — Blood samples and Nasosorption sampling
  Groups: Probable Idiopathic Pulmonary Fibrosis; Sarcoidosis,

SUMMARY:
The study will measure airway inflammation in probable idiopathic pulmonary fibrosis (IPF) and sarcoidosis as well as in healthy volunteers. This can help understand the molecular basis of these diseases, why these diseases happen, and what makes patients develop lung fibrosis. These insights should one day help to monitor patients and aid in their diagnosis and treatment.

DETAILED DESCRIPTION:
IPF is a progressive disease caused by irreversible scarring of the lung, and disease trajectory is not easily predicted based on clinical measurements. Biomarkers reflective of molecular pathways involved in IPF may help inform patient trajectory, but have been difficult to identify in circulation due to the disease manifesting in the lung. The study team will measure biomarkers from Probable IPF patients, sarcoidosis patients, and healthy volunteers using novel sampling methods involving absorption of upper and lower airway fluids. These novel sampling methods may enable less invasive and potentially more sensitive methods to detect disease activity and will be performed in IPF and sarcoidosis patients during a routine bronchoscopy procedure. The study team will compare the levels of biomarkers that have been shown to be predictive of disease course in airway fluids of probable IPF patients versus sarcoidosis and healthy controls. This study may help understand the molecular basis of IPF, and improve the understanding of diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Probable Idiopathic Pulmonary Fibrosis (IPF)
* Adult male or female patients aged 40 to 85 years
* Women of childbearing age should not be pregnant, planning to get pregnant or breast-feeding.
* Command of the English language to be able to give informed consent.
* Probable IPF requiring bronchoscopy to confirm the diagnosis, agreed within the local multi-disciplinary team (MDT).,according to the American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/ American Latin Thoracic Association (ATS/ERS/JRS/ALAT) guidelines (2018) (3)
* IPF disease diagnosis within the past 5 years
* Usual Interstitial Pneumonia (UIP) on HRCT scan.
* Recent lung function criteria:

  * Forced vital capacity (FVC) >40% of predicted value.
  * Carbon monoxide diffusing lung capacity (DLco) corrected for haemoglobin >30% of predicted value

Inclusion criteria for Sarcoidosis

* Adult male or female patients aged 18 years and over
* Women of childbearing age should not be pregnant, planning to get pregnant or breast-feeding.
* Clinical symptoms, CT scan and biopsy diagnosis of sarcoidosis
* Patients with lung parenchymal disease and pulmonary stage II or more
* Recent lung function criteria

  * FVC>50% predicted
  * DLCO >40% predicted

Inclusion criteria for Healthy Volunteers

* Age between 40 to 85 years, age and sex to match the group with IPF
* Healthy subjects without any diseases that may cause inflammation
* Women of childbearing age should not be pregnant, planning to get pregnant or breast-feeding.
* Currently non-smokers: see exclusion criteria

Exclusion Criteria:Exclusion Criteria for probable IPF and Sarcoidosis Patients

Respiratory Conditions other than IPF or sarcoidosis:

* Confirmed diagnosis of occupational lung disease
* Drug-induced lung disease or hypersensitivity pneumonitis
* Lung and systemic autoimmune disease including connective tissue disease. Patients with an auto-immune profile considered diagnostic for a specific connective tissue disease will be excluded, even in the absence of systemic symptoms. Non-specific rises in auto antibodies e.g. rheumatoid factor; anti-nuclear antibody etc. will not be used to exclude individuals from the study.
* Asbestosis or other asbestos related disease (pleural plaques, mesothelioma, asbestos pleural effusions)
* Granulomatous lung disease.
* Pulmonary artery hypertension (PAH) requiring a specific treatment.
* Predominant chronic obstructive pulmonary disease (COPD) with forced expiratory volume in 1 second /forced vital capacity (FEV1/FVC) <0.70.
* Patients with active tuberculosis or incompletely treated latent tuberculosis infection
* Lung cancer
* Upper respiratory tract infections in the past 6 weeks.

Systemic Conditions

* History of vasculitis, autoimmune or connective tissue disease
* Known human immunodeficiency virus (HIV) or chronic viral hepatitis
* Clinically significant diseases (other than IPF or sarcoidosis) that may alter respiratory biomarkers: including other respiratory, gastrointestinal, endocrine, haematological, cardiovascular, genitourinary, skin or neurological diseases.
* Recent or ongoing malignant diseases.
* Significant nasal anatomical defects preventing nasal sampling: including hypertrophy of turbinates, major septum deviation, nasal polyposis or recurrent sinusitis and nasal mucosal defects

Bronchoscopy Contraindications

Any contra-indication to bronchoscopy as set out in British Thoracic Society guidelines (34)

Smoking

A detailed smoking history will be taken from all participants: to include total pack years, smoking in the past year, and smoking in the past 2 weeks.

The history will include cigarettes, pipe smoking, cigars, vaping, and shisha. Any form of smoking is not permitted within 2 weeks of bronchoscopy.

5.4.2 Exclusion Criteria for Healthy Volunteers

* Current inflammatory/ immunological conditions. Any clinically significant diseases that may alter respiratory biomarkers: including respiratory, gastrointestinal, endocrine, haematological, cardiovascular, genitourinary, skin or neurological diseases.
* Recent or ongoing malignant diseases.
* Significant nasal anatomical defects preventing nasal sampling: including hypertrophy of turbinates, major septum deviation, nasal polyposis or recurrent sinusitis and nasal mucosal defects
* Upper respiratory tract infections in the past 6 weeks.
* Cigarette smoking:

no cigarettes in the last 2 weeks not more than 10 cigarettes in the past year <10 year lifetime pack history of smoking

-

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with probable IPF and Sarcoidosis will be included. Patients with probable IPF and Sarcoidosis will be selected from clinic lists for patients undergoing bronchoscopy as part of their clinical assessment, and they will be invited to participate in this study that involves additional sampling for clinical research purposes.
  Probable IPF patients must have Usual Interstitial Pneumonitis (UIP) on CT scan and will be sub classified by gas transfer (DLco corrected for haemoglobin as detailed below;
  * Mild (DLco>60)
  * Moderate (DLco 40-60)
  * Severe (DLco<40)
  Healthy volunteers (age/sex matched, non-smoking, without a clinical history of atopy).
  The patient populations will include:
  * Probable Idiopathic Pulmonary Fibrosis (IPF), n=30
  * Sarcoidosis patients, n=15
  * Healthy Volunteers n=15
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Levels of the of biomarker/mediator surfactant protein D (SPD) in bronchial Lining fluid in IPF and sarcoidosis patients | Baseline Bronchoscopy visit
  Comparisons will be made of bronchial lining fluid levels of biomarker/mediator surfactant protein D (SPD), in patients with IPF and sarcoidosis.
Levels of the biomarker/mediator CCL18 in bronchial Lining fluid in IPF and sarcoidosis patients. | Baseline Bronchoscopy visit
  Comparisons will be made of bronchial lining fluid levels of biomarker/mediator CCL18 in patients with IPF and sarcoidosis
Levels of the biomarker/mediator CXCL13 in bronchial Lining fluid in IPF and sarcoidosis patients. | Baseline Bronchoscopy visit
  Comparisons will be made of bronchial lining fluid levels of biomarker/mediator CXCL13 in patients with IPF and sarcoidosis.
Levels of the of biomarker/mediator periostin in bronchial Lining fluid in IPF and sarcoidosis patients. | Baseline Bronchoscopy visit
  Comparisons will be made of bronchial lining fluid levels of biomarker/mediator periostin in patients with IPF and sarcoidosis.

SECONDARY OUTCOMES:
Levels of Periostin in nasosorption samples within and across the 3 groups of participants | Through study completion, an average of 1 year
  Comparisons will be made of airways levels of biomarker/mediator periostin between patients with IPF and sarcoidosis and health volunteers.
Levels of surfactant protein (SPD) in nasosorption samples within and across the 3 groups | Through study completion, an average of 1 year
  Comparisons will be made of airways levels of biomarker/mediator surfactant protein D (SPD) between patients with IPF and sarcoidosis and health volunteers.
Levels of CCL18 in nasosorption samples within and across the 3 groups | Through study completion, an average of 1 year
  Comparisons will be made of airways levels of biomarker/mediator CCL18 between patients with IPF and sarcoidosis and health volunteers.
Levels of CXCL13 in nasosorption samples within and across the 3 groups | Through study completion, an average of 1 year
  Comparisons will be made of airways levels of biomarker/mediator CXCL13 between patients with IPF and sarcoidosis and health volunteers.
Levels of periostin in blood within and across the 3 groups of participants | Through study completion, an average of 1 year
  Comparison will be made of periostin levels in blood with nasosorption and bronchosorption levels across the 3 participant groups.
Levels of surfactant protein D (SPD in blood within and across the 3 groups of participants | Through study completion, an average of 1 year
  Comparison will be made of surfactant protein D (SPD levels in blood with nasosorption and bronchosorption levels across the 3 participant groups
Levels of CCL18 in blood within and across the 3 groups of participants | Through study completion, an average of 1 year
  Comparison will be made of CCL18 levels in blood with nasosorption and bronchosorption levels across the 3 participant groups.
Levels of CXCL13 in blood within and across the 3 groups of participants | Through study completion, an average of 1 year
  Comparison will be made of CXCL13 levels in blood with nasosorption and bronchosorption levels across the 3 participant groups.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Wickremasinghe, Principal Investigator — Physician

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT04494334/Prot_SAP_000.pdf